CLINICAL TRIAL: NCT05017350
Title: Hemostasis Using Radiofrequency Ablation for Track Bleeding After Liver Biopsy
Brief Title: Hemostasis Using Radiofrequency Ablation for Track Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyoung Doo Song (Other)
Responsible Party: Sponsor-Investigator, Kyoung Doo Song, Associate Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-04-028-003
Record Dates: First submitted 2021-08-03; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Bleeding
Keywords: liver; track bleeding; radiofrequency ablation
MeSH Terms: conditions — Hemorrhage | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiofrequency ablation group (Experimental): hemostasis using radiofrequency ablation for track bleeding
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: radiofrequency ablation — Under the ultrasound guidance, the electrode is inserted into the bleeding focus of the liver and the bleeding focus is ablated.

SUMMARY:
This study aims to evaluate the usefulness of hemostasis using radiofrequency ablation for track bleeding that has occurred after percutaneous biopsy of the liver.

DETAILED DESCRIPTION:
Purpose: To evaluate the usefulness of hemostasis using radiofrequency ablation for track bleeding after percutaneous liver biopsy.

Method:

* Enroll patients who continue to bleed despite conservative treatment for track bleeding that has occurred after liver biopsy.
* Radiofreqeuncy ablation: Under monitoring vital signs and controlling pain with intravenous agents, the electrode is inserted into the bleeding focus. The bleeding focus is ablated.
* Hemostasis is evaluated by ultrasound (right after radiofrequency ablation), CT scan (after the radiofrequency ablation), and ultrasound (the day after radiofrequency ablation)
* If hemostasis fails using radiofrequency ablation, transarterial hepatic embolization is performed immediately.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound guided percutaneous liver biopsy at Samsung Medical Center
* Track bleeding after biopsy
* Persistent track bleeding even after conservative management
* Consent to this study

Exclusion Criteria:

* Not consent to this study
* <20 years old or >=80 years old
* Contraindication to radiofrequency ablation
* Radiofrequency ablation for track bleeding is not technically possible.
* Unstable vital signs

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
hemostasis rate | immediately after radiofrequency ablation
  success rate of hemostasis using radiofrequency ablation on CT taken after radiofrequency ablation

SECONDARY OUTCOMES:
complication rate | immediately after radiofrequency ablation
  complication rate associated with radiofrequency ablation on CT taken after radiofrequency ablation

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Doo Song, Professor, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No